CLINICAL TRIAL: NCT03549702
Title: Subcutaneous Tissue Irrigation With Povidone Iodine in Decreasing the Rate of Surgical Site Infection Following Cesarean Section (Randomized Control Trial)
Brief Title: Subcutaneous Tissue Irrigation With Povidone Iodine in Decreasing the Rate of Surgical Site Infection Following Cesarean Section
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, George Adel Azmy, Specialist in Obstetrics and Gynecology, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PovidIodCS
Record Dates: First submitted 2018-03-09; First posted 2018-06-08 (Actual); Last update posted 2018-06-08 (Actual); Status verified 2018-05

CONDITIONS: Surgical Site Infection
MeSH Terms: conditions — Surgical Wound Infection | interventions — Povidone-Iodine; Solutions

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Povidone irrigation Group (Active Comparator): Includes the 100 women who will undergo elective caesarian section with subcutaneous tissue irrigation with Povidone iodine 1% solution.
  Interventions: Drug: Povidone iodine 1% solution
- Control Group (No Intervention): Includes the 100 women who will undergo elective caesarian section without subcutaneous tissue irrigation with Povidone iodine 1% solution.

INTERVENTIONS:
Drug: Povidone iodine 1% solution — irrigation of subcutaneous tissue with Povidone-Iodine prior to skin closure
  Arms: Povidone irrigation Group

SUMMARY:
This study aims to assess the efficacy of Povidone Iodine (Betadine®) irrigation of subcutaneous tissue prior to skin closure in reducing the incidence of surgical site infection after elective caesarean section and post discharge.

DETAILED DESCRIPTION:
All women will be counseled regarding mode of intervention and informed consent will be obtained. All women will be subjected to complete history taking, routine antenatal examination and investigations especially Hemoglobin test and 2 hour glucose tolerance test, treatment of genital or urinary tract infections if diagnosed. Routine obstetric ultrasound examination.

Primary Outcome :

Surgical site infection up to 14 days following elective caesarian section.

Criteria of Surgical site infection:

Infection involves only skin and subcutaneous tissue of this incision. Occurs within 14 days after the operative procedure.

Includes at least one of the following:

1. purulent drainage is present (culture documentation not required)
2. organisms are isolated from fluid/tissue of the superficial incision
3. at least one sign of inflammation (eg, pain or tenderness, induration, erythema, local warmth of the wound) is present.
4. the wound is deliberately opened by the surgeon
5. the surgeon or clinician declares the wound infected.

Secondary Outcome :

1. The need for secondary sutures closure of the infected wound after cleaning and debridement.
2. The need for other doses of antibiotic rather than the preoperative prophylactic one.
3. Postoperative fever exceeding 38.2, 24 hours following the caesarian section after exclusion of the other possible causes (eg: DVT, chest infections, Urinary tract infections).
4. The duration of post operative hospital stay
5. Coast effectiveness of hospital stay duration.

Randomization :

The study population will be randomly distributed according to the mode of intervention into 2 groups.

Randomization is performed using a Computer generated randomization system. Table of randomization is obtained.

Group 1 Includes the 100 women who will undergo elective caesarian section with subcutaneous tissue irrigation with Povidone iodine 1% solution.

Nature of Povidone Iodine: It's a stable chemical complex of polyvinylpyrrolidone and elemental iodine.with chemical formula (C6H9I2NO).

Antiseptic properties: it's a broad spectrum antiseptic for topical application in the treatment and prevention of infection in wounds, using the antiseptic properties of iodine.

Iodine has been recognized as an effective broad-spectrum bactericide, and is also effective against yeasts, molds, fungi, viruses, and protozoans.

In addition, it has been demonstrated that bacteria do not develop resistance to Povidone Iodine (Fleischer and Reimer, 1997).

Prophylactic 1gm of 3rd generation cephalosporins 30 minutes prior to skin incision.

The level of surgeon will be 2nd year residency or higher. Skin incision will be done by scalpel in Pfannenstiel manner. Subcutaneous tissue incision and division will be done using scalpel. Rectus sheath division will be done by scalpel with good hemostasis. Opening of the parietal peritoneum either sharp or blunt. Opening of the uterus in a C-shaped manner. Oxytocin 5 IU by slow intravenous injection will be used to encourage contraction of the uterus and to decrease blood loss.

The placenta will be removed using controlled cord traction and not manual removal.

Closure of the uterus in two continuous layers using polyglactin 910 No 1. Closure of parietal peritoneal. Closure of the rectus sheath in a continuous fashion using polyglactin 910 No1. Good hemostasis of subcutaneous tissue using the diathermy in coagulation mood. Irrigation of the subcutaneous tissue layers using povidone iodine using Betadine filled 20 cm syringe.

No insertion of subcutaneous tissue drain. No interrupted sutures in the skin. Approximating of the subcutaneous tissue using polyglactin 910 (2-0) if the tissue thickness more than 2 cm .

Closure of the skin using polypropylene (2-0) in subcuticular manner.

Group 2:

Includes the 100 women who will undergo elective caesarian section without subcutaneous tissue irrigation with Povidone iodine 1% solution.

Same steps as group 1 without subcutaneous tissue irrigation with Povidone iodine.

Allocation and Concealment 200 eligible women (who fulfill the inclusion and exclusion criteria) are to be randomly allocated into one of the two groups. Concealed allocation is adopted, however, in order to minimize selection bias. The allocated group numbers are concealed in serially-numbered opaque envelopes. Each envelope will contain the number of one of the two arms of the study, envelopes will be put in a box, and each woman under the study will pick one envelope which corresponds to the group to which she will be allocated. The envelopes are unsealed after recruitment of the cases.

ELIGIBILITY:
Inclusion Criteria:

1. Age: from 20 to 35 old years.
2. Elective cesarean section.
3. Caesarean section time from skin incision to skin closure less than 60 minutes.
4. Preoperative Hemoglobin more than 10 gm /dl.
5. Body Mass Index: 20_30 Kg/m2 .

Exclusion Criteria:

1. Body Mass Index: <20 or >30 Kg/m2.
2. Diabetic patient.
3. Feverish patient.
4. Patient using steroids for chronic illness.
5. Hypertension chronic or with pregnancy.
6. Prelabour rupture of membranes.
7. Difference in pre and postoperative hemoglobin more than 10%.
8. Patients have a Coagulopathy disorder.
9. Multiple pregnancy.

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2018-02-28 (Actual); Study Completion 2018-03-03 (Actual)

PRIMARY OUTCOMES:
Surgical site infection up to 14 days following elective caesarian section. | 14 Days
  * Infection involves only skin and subcutaneous tissue of this incision.
  * Occurs within 14 days after the operative procedure.
  * Includes at least one of the following:
    1. purulent drainage is present (culture documentation not required)
    2. organisms are isolated from fluid/tissue of the superficial incision
    3. at least one sign of inflammation (eg, pain or tenderness, induration, erythema, local warmth of the wound) is present.
    4. the wound is deliberately opened by the surgeon
    5. the surgeon or clinician declares the wound infected.

CONTACTS AND LOCATIONS:
Overall Officials: George Azmy, MBBCH, Principal Investigator — Specialist of Obstetrics and Gynecology
Locations (1):
- Faculty of Medicine - Ain SHams University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided